CLINICAL TRIAL: NCT03413436
Title: Multicenter Comparative of Toxicity and Effectiveness of Lobaplation or Cisplatin Based Adjuvant Chemotherapy in Esophageal Carcinoma
Brief Title: Lobaplation or Cisplatin in Adjuvant Chemotherapy for Esophageal Carcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH1801
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Esophageal Cancer
Keywords: adjuvant chemotherapy; multicenter retrospective study
MeSH Terms: conditions — Esophageal Neoplasms | interventions — lobaplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lobaplatin group (Experimental): i) thoracic ESCC stage II to III; ii) without any preoperation treatment for ESCC; iii) underwent R0 resection; iv) received at least one cycle ajuvant chemotherapy of Lobaplatin plus Docetaxel; v) without ajuvant radiotherapy/chemoradiotherapy; vi) without history of other type of cancer. Completed clinical, pathological and follow up data.
  Interventions: Drug: Lobaplatin
- Cisplatin group (Active Comparator): i) thoracic ESCC stage II to III; ii) without any preoperation treatment for ESCC; iii) underwent R0 resection; iv) received at least one cycle ajuvant chemotherapy of Cisplatin plus Docetaxel; v) without ajuvant radiotherapy/chemoradiotherapy; vi) without history of other type of cancer. Completed clinical, pathological and follow up data.
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Lobaplatin — at least one cycle adjuvant chemotherapy after esophagectomy
  Arms: Lobaplatin group
Drug: Cisplatin — at least one cycle adjuvant chemotherapy after esophagectomy
  Arms: Cisplatin group

SUMMARY:
The multicenter real-world and propensity score matching comparative study was designed to explore the toxicity and effectiveness of Lobaplation or Cisplatin based adjuvant chemotherapy in esophageal carcinoma

DETAILED DESCRIPTION:
This trial is a multicenter real-world retrospective comparative study. The patients with thoracic esophageal squamous cell carcinoma, esophagectomy and adjuvant chemotherapy(Cisplatin plus Docetaxel or Lobaplatin plus Docetaxel) from 6 centers in China were enrolled from Jan.2013 to Dec.2016. Completed clinical and pathological data were collected from Large-scale Data Analysis Center of Cancer Precision Medicine-LinkDoc database and analyzed by using data technology support from LinkDoc by using R-language. A hybrid solution for extracting structured medical infromation from unstructured data in medical records via a double-reading/entry system. The World Health Organization (Toxicity Grading Scale for Determining the Severity of Adverse Events) was used. The side effects of adjuvant chemotherapy and overall survival rate were compared by a propensity score. The 6 centers are The affiliated Cancer Hospital of ZhengZhou university/Henan Cancer Hospital, Anyang Cancer Hospital, Anhui Province Hospital, The first affiliated Hospital of Anhui university, Tangdu Hospital/the affiliated Hospital of Fourth Military Medical University, The First Affiliated Hospital of Xi'an Jiao Tong University.

ELIGIBILITY:
Inclusion Criteria:

* i) thoracic ESCC stage II to III; ii) without any preoperation treatment for ESCC; iii) underwent R0 resection; iv) received ajuvant chemotherapy of Cisplatin plus Docetaxel or Lobaplatin plus Docetaxel.

Exclusion Criteria:

* i) with ajuvant radiotherapy/chemoradiotherapy; ii) history of other type of cancer iii) without completed clinical, pathological and follow up data.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 733 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years
  The days from esophagectomy to cancer specific death

SECONDARY OUTCOMES:
toxicities of adjuvant chemotherapy | from chemotherapy to 3 month after last cycle adjuvant chemotherapy
  According to National Cancer Institute Common Terminology Criteria for Adverse Event,Version 3.0(CTC AE3.0).

CONTACTS AND LOCATIONS:
Overall Officials: Yin Li, Dr., Principal Investigator — The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China

REFERENCES:
- [Derived] Zheng Y, Li Y, Liu X, Sun H, Liang G, Hu J, Li L, Xing W. Multicentre Comparison of the Toxicity and Effectiveness of Lobaplatin-Based Versus Cisplatin-Based Adjuvant Chemotherapy in Oesophageal Carcinoma. Front Oncol. 2021 Sep 13;11:668140. doi: 10.3389/fonc.2021.668140. eCollection 2021. PMID 34589419